CLINICAL TRIAL: NCT00158990
Title: Triiodothyronine (T3) Supplementation in Bipolar and Unipolar Depression: A Random Assignment, Double Blind, Placebo-Controlled Study.
Brief Title: Triiodothyronine (T3) Supplementation in the Treatment of Bipolar and Unipolar Depression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPL-0100-HMO-CTIL
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2005-08

CONDITIONS: Major Depression; Bipolar Disorder; Unipolar Depression
Keywords: major depression; bipolar disorder; unipolar depression; sertraline; triiodothyronine
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depressive Disorder | interventions — Triiodothyronine; Sertraline

INTERVENTIONS:
Drug: triiodothyronine
Drug: sertraline

SUMMARY:
The purpose of this project is to determine whether concurrent treatment of patients with major depression (unipolar or bipolar) with triiodothyronine (T3) and sertraline, will lead to a stronger and/or more rapid antidepressant effect than treatment with sertraline alone.

DETAILED DESCRIPTION:
AIM: To determine the therapeutic efficacy and adverse effects of triiodothyronine (T3) as a supplement to the treatment of bipolar depression (BPD) with a mood stabilizer (MS) (lithium - Li, valproic acid - VPA or carbamazepine - CBZ) and the specific serotonin reuptake inhibitor (SSRI), sertraline; and as a supplement to the treatment of unipolar depression (UPD) with sertraline.

METHOD: A random assignment, double blind, placebo-controlled trial separately evaluating patients with a) BPD who are treated with MS + sertraline + T3 or MS + sertraline + placebo and b) UPD who are treated with sertraline + T3 or sertraline + placebo, for up to 8 weeks in both cases. The design of the trial will permit both the outcome of treatment and the speed of response to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Major Depressive Episode (MDE) in the context of Bipolar Disorder I or II (BPD-I or BPD-II) or Major Depressive Disorder (UPD), according to DSM-IV criteria, without psychotic features.
2. Hamilton Depression Scale (HAM-D) total >16 with item 1 (depressed mood) >2.
3. Age 18-70 years, male or female.
4. Competent and willing to give written informed consent.

Exclusion Criteria:

1. No clinical hyper- or hypothyroidism nor other thyroid illness.
2. No neurological or other physical illness that may impact upon the study or limit prescription of the study medications.
3. No lifetime history of substance or alcohol dependence or of abuse in the preceding 12 months.
4. No significant suicidal risk (HAM-D item 3 (suicide) <3).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2002-10; Study Completion 2007-07

PRIMARY OUTCOMES:
Response - HAM-D-21 improvement >50% at 8 weeks
Remission - final HAM-D-21 total <7 at 8 weeks

SECONDARY OUTCOMES:
Rate of change in HAM-D-21 scores over 8 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Lerer, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Global Medical Institutes, Princeton, New Jersey, United States
- Hadassah Medical Organisation, Jerusalem, Israel

REFERENCES:
- [Derived] Cooper-Kazaz R, Apter JT, Cohen R, Karagichev L, Muhammed-Moussa S, Grupper D, Drori T, Newman ME, Sackeim HA, Glaser B, Lerer B. Combined treatment with sertraline and liothyronine in major depression: a randomized, double-blind, placebo-controlled trial. Arch Gen Psychiatry. 2007 Jun;64(6):679-88. doi: 10.1001/archpsyc.64.6.679. PMID 17548749